CLINICAL TRIAL: NCT00998010
Title: Phase II Trial of Velcade (Bortezomib) in Combination With Temozolomide and Regional Radiation Therapy for Upfront Treatment of Patients With Newly-diagnosed Glioblastoma Multiforme
Brief Title: Bortezomib, Temozolomide, and Regional Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme or Gliosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-002222; UCLA-X05303; CDR0000657015; MILLENNIUM-UCLA-X05303; 09-03-084 (Other: UCLA IRB)
Record Dates: First submitted 2009-10-17; First posted 2009-10-20 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2019-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Patients receive bortezomib IV on days 1, 4, 8, 11, 29, 32, 36, and 39 and oral temozolomide on days 1-42.Patients undergo external-beam fractionated regional radiotherapy 5 days a week for 6 weeks in the absence of disease progression or unacceptable toxicity.2-6 weeks after radiotherapy, patients receive bortezomib IV on days 1, 4, 8, and 11 and oral temozolomide on days 1-5.Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib + temozolomide+ radiation therapy

INTERVENTIONS:
Drug: bortezomib + temozolomide+ radiation therapy — Patients will be treated with Bortezomib at 1.3 mg/m2 IV on days1,4,8,11,29,32,36 and 39 and Temozolomide on 75mg/m2 daily during radiation. External beam fractionated regional radiation will be given on consecutive week days at 200 centigray (cGy) daily doses to a total dose of 6000 cGy.

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving bortezomib together with temozolomide and radiation therapy may kill more tumor cells and allow doctors to save the part of the body where the cancer started.

PURPOSE: This phase II trial is studying the side effects and how well bortezomib works when given together with temozolomide and regional radiation therapy in treating patients with newly diagnosed glioblastoma multiforme or gliosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the overall survival at 2 years of patients with newly diagnosed glioblastoma multiforme treated with bortezomib in combination with temozolomide and regional radiotherapy followed by maintenance therapy comprising bortezomib and temozolomide.

Secondary

* Investigate further the safety and tolerability of this regimen in these patients.
* Determine the molecular characterization of tumor tissue and correlate these findings with response.

OUTLINE: This is a multicenter study.

* Adjuvant chemotherapy: Patients receive bortezomib IV on days 1, 4, 8, 11, 29, 32, 36, and 39 and oral temozolomide on days 1-42. Patients undergo external-beam fractionated regional radiotherapy 5 days a week for 6 weeks in the absence of disease progression or unacceptable toxicity.
* Maintenance: Beginning 2-6 weeks after radiotherapy, patients receive bortezomib IV on days 1, 4, 8, and 11 and oral temozolomide on days 1-5. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

Tumor tissue samples are collected at baseline (from surgery) and periodically during study for further analysis.

After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Must be >- 18 years old, with a life expectancy > 8 weeks
* Histologically confirmed intracranial glioblastoma multiforme (GBM) or gliosarcoma
* Must submit an unstained paraffin block or slides from surgical procedure
* Patients without prior treatment and with prior diagnosis of lower-grade gliomas that have been upgraded to GBM after repeated resection allowed
* At least 21 days since cranial MRI or contrast CT scan OR ≥ 96 hours since cranial MRI or contrast CT scan for patients who underwent surgical resection
* Measurable or assessable disease
* Voluntary written informed consent obtained before performance of any study related procedure not part of normal medical care.
* Karnofsky performance status > 60%
* White Blood Count (WBC) ≥ 3,000/mm^3
* absoulte neutrophil count(ANC) ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* Bilirubin < 2.5 times upper limit of normal (ULN)
* serum glutamic-oxaloacetic transaminase (SGOT) < 2.5 times ULN
* Creatinine < 1.5 mg/dL
* Creatinine clearance ≥ 20 mL/minute
* Serum sodium > 130 mmol/L
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients on Enzyme-Inducing Antiepileptic Drugs (EIAED) must be transitioned to non- EAIED for ≥ 2 weeks
* Concurrent full-dose warfarin or its equivalent (e.g., unfractionated and/or low molecular weight heparin) allowed

Exclusion Criteria:

* peripheral neuropathy ≥ grade 2
* Myocardial infarction within the past 6 months
* New York Heart Association (NYHA) class III or IV heart failure
* Uncontrolled angina
* Severe uncontrolled ventricular arrhythmias
* Electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* hypersensitivity to bortezomib, boron, or mannitol
* serious medical or psychiatric illness that would interfere with study participation including, but not limited to, any of the following:
* Ongoing or active infection requiring IV antibiotics
* Psychiatric illness and/or social situations that would limit compliance with study requirements
* Disorders associated with a significant immunocompromised state (e.g., HIV, systemic lupus erythematosus)
* history of stroke within the past 6 months
* other malignancy within the past 3 years except completely resected basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy (i.e., cervical cancer), or low-risk prostate cancer after curative therapy
* significant medical illness that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* disease that will obscure toxicity or dangerously alter drug metabolism
* viral hepatitis (HBV surface antigen positive) or active hepatitis C infection
* Prior or concurrent corticosteroids, automated external defibrillator, analgesics, and other drugs to treat symptoms or prevent complications allowed
* concurrent investigational drugs that must be stopped at least 4 months prior to therapy.
* prior radiotherapy to the brain
* prior cytotoxic or noncytotoxic drug therapy or experimental drug therapy (including chemotherapy, hormonal therapy, or immunotherapy) directed against the brain tumor
* prior polifeprosan 20 with carmustine implant (Gliadel wafer)
* concurrent stereotactic radiosurgery or brachytherapy
* concurrent sargramostim
* concurrent inducers of CYP450 3A4 (e.g., enzyme-inducing anti-epileptic drugs [EIAED])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10-03 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lai, MD, PhD, Principal Investigator — Ronald Reagan UCLA Medical Center
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 10/03/2011 - 4/17/2015 Location: University of California at Los Angeles, Columbia University, New York.
Pre-assignment Details: There are no pre-assignment details to describe.
Period: Overall Study
Arm/Group | Experimental
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Twenty-four patients with newly diagnosed Glioblastoma Multiforme were enrolled in this study
Groups:
- Experimental: Patients receive bortezomib IV on days 1, 4, 8, 11, 29, 32, 36, and 39 and oral temozolomide on days 1-42.Patients undergo external-beam fractionated regional radiotherapy 5 days a week for 6 weeks in the absence of disease progression or unacceptable toxicity.2-6 weeks after radiotherapy, patients receive bortezomib IV on days 1, 4, 8, and 11 and oral temozolomide on days 1-5.Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  bortezomib + temozolomide+ radiation therapy: Patients will be treated with Bortezomib at 1.3 mg/m2 IV on days1,4,8,11,29,32,36 and 39 and Temozolomide on 75mg/m2 daily during radiation. External beam fractionated regional radiation will be given on consecutive week days at 200 centigrays (cGy) daily doses to a total dose of 6000 cGy.
Arm/Group | Experimental
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years]
  Age Range | 57 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Estimate the overall survival in subjects with newly-diagnosed glioblastoma (GBM) treated with bortezomib/temozolomide/radiation followed by bortezomib/temozolomide for 24 cycles until progression is detected or for up to 24 cycles (~2 years).
Time Frame: 2 years
Population: From completion of radiation treatment to tumor progression
Measure: Mean (95% Confidence Interval); unit: months
Groups:
- Experimental: Patients receive bortezomib IV on days 1, 4, 8, 11, 29, 32, 36, and 39 and oral temozolomide on days 1-42.Patients undergo external-beam fractionated regional radiotherapy 5 days a week for 6 weeks in the absence of disease progression or unacceptable toxicity.2-6 weeks after radiotherapy, patients receive bortezomib IV on days 1, 4, 8, and 11 and oral temozolomide on days 1-5.Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  bortezomib + temozolomide+ radiation therapy: Patients will be treated with Bortezomib at 1.3 mg/m2 IV on days1,4,8,11,29,32,36 and 39 and Temozolomide on 75mg/m2 daily during radiation. External beam fractionated regional radiation will be given on consecutive week days at 200cGy daily doses to a total dose of 6000 cGy.
Arm/Group | Experimental
Number analyzed (Participants) | 24
months | 19.1 [6.7 to 31.4]

2. Secondary Outcome: Toxicity Assessed According to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 24
Participants
  Radiotherapy phase: Grade 3 toxicity | 6
  Radiotherapy phase: Grade 4 Toxicity | 1
  Radiotherapy phase: < Grade 3 Toxicity | 17
  Post Radiotherapy phase: Grade 3 toxicity | 7
  Post Radiotherapy phase: Grade 4 Toxicity | 0
  Post Radiotherapy phase: < Grade 3 Toxicity | 17
  Follow-up phase: Grade 3 toxicity | 0
  Follow-up phase: Grade 4 Toxicity | 0
  Follow-up phase: < Grade 3 Toxicity | 24

3. Secondary Outcome: Time to Progression
Description: Median time to tumor progression. Because many newly-diagnosed patients are likely not to have evaluable disease due to gross total resections. A 7-point scale was used to guide Magnetic resonance imaging (MRI) assessment to determine progression in this study. A -2 or -3 assessment will be taken as progression.
  The 7-point scale is listed below. complete resolution of tumor: 3 tumor definitely smaller: 2 tumor probably smaller: 1 tumor unchanged: 0 tumor probably worse: -1 tumor definitely worse: -2 new lesion: -3
Time Frame: From the completion of radiation treatment to tumor progression
Population: From the completion of radiation treatment to tumor progression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 24
months | 6.2 [3.7 to 8.8]

4. Secondary Outcome: Survival at 1 Year
Description: Overall Survival at 12 months from completion of radiation treatment
Time Frame: 1 year
Population: 12 months from completion of radiation treatment to tumor progression.
Measure: Median (Full Range); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 24
percentage of participants | 87.5 [66.1 to 95.8]

5. Secondary Outcome: Tumor Progression as Assessed by Magnetic Resonance Imaging (MRI) and Neurologic Exam
Description: MRI will be done 2 weeks after completion of radiation and then every 8 weeks. Neurologic exam to be performed every 2 weeks during radiation therapy, then every every 4 weeks after radiation is completed.
Time Frame: at 6, 12, 18 and 24 months from completion of radiation treatment.
Population: Outcome was not analyzed separately, MRI and Neurological exam were to determine the progression status, and finally reflected as Progression Free Survival and Overall Survival
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 24
percentage of participants
  Progression Free Survival rate at 6 months | 54.2 [32.7 to 71.4]
  Progression Free Survival rate at 12 months | 29.2 [13.0 to 47.6]
  Progression Free Survival rate at 18 months | 25.0 [10.2 to 43.1]
  Progression Free Survival rate at 24 moths | 25 [10.2 to 43.1]

ADVERSE EVENTS:
Time Frame: Adverse Events data was collected up to 2 years from the completion of radiation treatment
Description: Systemic adverse event assessment occurred weekly during radiation treatment period, and on Day 1 and Day 21 of each 28-day maintenance treatment cycle, and within 30 days after administration of the last dost of study drug bortezomib.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 15/24
Serious Adverse Events (participants affected / at risk) | 5/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=24)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Shingles (Infections and infestations) | 1 (1) — varicella-zoster virus (VZV) Infection
Hydrocephalus (Nervous system disorders) | 1 (1) — Ventriculoperitoneal (VP) Shunt placement
Craniotomy (Nervous system disorders) | 1 (1) — Craniotomy due to PD
Pullmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hydrocephalus placement
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=24)
Anemia (Blood and lymphatic system disorders) | 9 (36)
Leukocytopenia (Blood and lymphatic system disorders) | 9 (44)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (10)
Neutropenia (Blood and lymphatic system disorders) | 6 (30)
lymphopenia (Blood and lymphatic system disorders) | 14 (107)
Encephalopathy (elevated ammonia) (Nervous system disorders) | 1 (1)
Vasogenic edema (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 17 (21)
Fever (General disorders) | 4 (5)
Malaise (General disorders) | 1 (2)
Weight Loss (General disorders) | 3 (3)
Weight gain (General disorders) | 4 (4)
Insomnia (General disorders) | 4 (4)
Hypersomnia (General disorders) | 1 (1)
Chills (General disorders) | 3 (4)
Increased appetite (General disorders) | 2 (2)
Injection site reaction (Skin and subcutaneous tissue disorders) | 13 (13)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2)
skin rash-Radiodermatitis (Skin and subcutaneous tissue disorders) | 4 (4)
Skin rash- diffuse (Skin and subcutaneous tissue disorders) | 3 (5)
Wound complication (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8)
Other-Blepharitis (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
other- Skin Tears L. Forearm L. Peritibial region (Skin and subcutaneous tissue disorders) | 1 (1)
skin rash-Periorbital (Skin and subcutaneous tissue disorders) | 1 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
skin rash (bactrim allergy) (Skin and subcutaneous tissue disorders) | 2 (3)
Skin Rash/acne (Skin and subcutaneous tissue disorders) | 2 (2)
bruising Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Cushingoid appearance (Endocrine disorders) | 2 (2)
Ocular/ chalazion (Eye disorders) | 2 (2)
Ocular/visual Xerophtalmia/dry eyes (Eye disorders) | 1 (1)
Ocular/visual Blurred vision (Eye disorders) | 1 (1)
Poor Appetite/anorexia (Gastrointestinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 11 (14)
Vomiting (Gastrointestinal disorders) | 6 (9)
Dehydration (Gastrointestinal disorders) | 1 (1)
Bloating/Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Cardiac/general Hypertension (Cardiac disorders) | 1 (1)
Cardiac/general Hypotension (Cardiac disorders) | 1 (1)
Cardiac arrhythmia Tachycardia (Cardiac disorders) | 2 (2)
Allergy/immunology Allergic rhinitis (nasal congestion ) (Immune system disorders) | 1 (1)
Other-Pelvic infection (Infections and infestations) | 1 (1)
Oral thrush (Infections and infestations) | 2 (2)
Ear Infection/otitis media (Infections and infestations) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2)
Stye on LL conjunctival border (Eye disorders) | 1 (1)
Other-Herpes zoster infection (Infections and infestations) | 2 (2)
Lymphatics Limb edema (Blood and lymphatic system disorders) | 3 (3)
Lymphatics/edema Swelling on the lips (Blood and lymphatic system disorders) | 1 (1)
Personality/behavioral change (Psychiatric disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Elevated bilirubin (Metabolism and nutrition disorders) | 4 (16)
Elevated ALP (Metabolism and nutrition disorders) | 1 (1)
Elevated ALT (Metabolism and nutrition disorders) | 5 (6)
Elevated AST (Metabolism and nutrition disorders) | 4 (5)
Elevated LDH (Metabolism and nutrition disorders) | 1 (2)
Hyperglicemia (Metabolism and nutrition disorders) | 4 (8)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4)
Elevated CREATINIE (Metabolism and nutrition disorders) | 1 (1)
Decrease GFR (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)
Elevated triglycerides (Metabolism and nutrition disorders) | 1 (1)
Cramping (Musculoskeletal and connective tissue disorders) | 2 (2)
meniscal tear (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Gait/Walking (Musculoskeletal and connective tissue disorders) | 3 (5)
Seizure (Nervous system disorders) | 5 (11)
Tremor (Nervous system disorders) | 2 (3)
Mood alteration (Nervous system disorders) | 6 (11)
Confusion (Nervous system disorders) | 5 (6)
Memory impairment (Nervous system disorders) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Motor neuropathy (Nervous system disorders) | 1 (1)
Sensory neuropathy (Nervous system disorders) | 4 (4)
Hydrocephalus (Nervous system disorders) | 2 (3)
Paresthesia (Nervous system disorders) | 3 (3)
Motor weakness (Nervous system disorders) | 3 (3)
Falls (Nervous system disorders) | 1 (1)
Positional Dizziness (Nervous system disorders) | 3 (3)
voice changes Dysarthria (Nervous system disorders) | 2 (2)
Alexia (Nervous system disorders) | 1 (1)
Lack of motivation (Nervous system disorders) | 1 (1)
Difficulty with concentration (Nervous system disorders) | 2 (2)
extrapyramidal involuntary Movement Restless legs (Nervous system disorders) | 1 (1)
other- Abulia (Nervous system disorders) | 1 (1)
Aphasia (Nervous system disorders) | 2 (2)
dysphagia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Olecranon bursitis (General disorders) | 1 (1)
Dental: periodontal disease-sensitivity (General disorders) | 1 (1)
Headache (Nervous system disorders) | 14 (23)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other-VZV infection related pain (General disorders) | 1 (1)
Cramping/Bilateral Lower Extremities (General disorders) | 1 (1)
Back (Musculoskeletal and connective tissue disorders) | 2 (2)
Nose (Musculoskeletal and connective tissue disorders) | 3 (3)
Dispnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
other-Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 3 (4)

LIMITATIONS AND CAVEATS:
Enrolls newly diagnosed GBM patient and requires collection of frozen and paraffin tumor tissue in all study patients from original surgery. Tissues for methylated (MGHT) and isocitrate dehydrogengenotyping and correlative molecular characterization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-02-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT00998010/Prot_SAP_000.pdf
  • Informed Consent Form (2015-01-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT00998010/ICF_001.pdf